CLINICAL TRIAL: NCT01071525
Title: The Effect of Niacin Administration on Oxidative Stress in Patients With Hypercholesterolmia, as Measured by the Use of a Novel Biomarker
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dr Shadi Hamoud, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Niacin-OS
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2010-03-01 (Estimated); Status verified 2010-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Niacin (Active Comparator): Hypercholesterolemic patients with high-density lipoprotein (HDL) less than 40 mg% will receive Niacin\Laropiprant.
  Interventions: Drug: Niacin\Laropiprant
- Control (No Intervention): Maching subjects will receive no medication, Blood tests will be drawn for laboratory tests.
  Interventions: Drug: Niacin\Laropiprant

INTERVENTIONS:
Drug: Niacin\Laropiprant — Hypercholesterolemic patients with low HDL will receive Niacin\Laropiprant

SUMMARY:
1. Treatment of Hypercholesterolemic patients with niacin will cause a significant decrease in oxidative stress and a decrease in the atherogenecity in blood samples of the patients.
2. A possible correlation between oxidative stress in hypercholesterolemic patients taking niacin to clinical hypercholesterolemia parameters is possible.
3. Using a novel biomarker will enable a precise detection of the change in the oxidative stress in hypercholesterolemic patients.

ELIGIBILITY:
Inclusion Criteria:

* Hypercholesterolemia,
* age above eighteen

Exclusion Criteria:

* Treatment with fibrates,
* Pregnant/Breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-08 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Effect on oxidative stress | three months

CONTACTS AND LOCATIONS:
Overall Officials: Liz Phima, Study Director — Study Coordinator
Locations (1):
- Rambam Health Care Campus, Haifa, Israel